CLINICAL TRIAL: NCT03608527
Title: The Impact of Motor Rehabilitation on the Dynamic Properties of the Brain: Towards the Individual Tailoring of Therapeutic Interventions in Multiple Sclerosis Patients
Brief Title: Adaptive Plasticity Following Rehabilitation in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Italiana Sclerosi Multipla (Other)
Collaborators: Universita degli Studi di Genova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FISM 2011R8
Record Dates: First submitted 2018-07-13; First posted 2018-08-01 (Actual); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Multiple Sclerosis
Keywords: Upper limb motor rehabilitation; Voluntary movements; functional magnetic resonance imaging
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active motor treatment (AMT) group (Experimental): 15 people with multiple sclerosis performing a 8 week rehabilitative treatment based on task-oriented voluntary exercises (3 sessions/week).
  Interventions: Behavioral: Voluntary-based upper limb motor rehabilitation
- Passive motor treatment (PMT) group (Active Comparator): 15 people with multiple sclerosis performing a 8 week passive mobilization delivered by a physical therapist (3 sessions/week).
  Interventions: Behavioral: Passive upper limb mobilization

INTERVENTIONS:
Behavioral: Voluntary-based upper limb motor rehabilitation — Exercises for neuromuscular control to improve proprioceptive sensibility, muscle strength, stability and coordination of the upper limbs, mainly including task-oriented movements with the goal to improve activities of daily living. Both proximal and distal muscles are involved, in actions such as grasping wooden cubes of different sizes, pinching, reaching targets displayed in front of the patient, and doing patchwork or paper mandala.
  Arms: Active motor treatment (AMT) group
Behavioral: Passive upper limb mobilization — Passive mobilization delivered by a physical therapist of shoulder, elbow, wrist and fingers without detectable muscle activity.
  Arms: Passive motor treatment (PMT) group

SUMMARY:
Motor learning can induce significant changes in the human brain through neural plasticity processes, which play a crucial role in the brain functional reorganization in response to external stimuli and/or to pathological conditions. For example, people with multiple sclerosis present motor deficits often associated with cerebral activity alteration. However, whether these brain activation changes contribute to or protect against motor performance deficits still needs to be determined.

Moreover, rehabilitation protocols could be designed to obtain efficient brain adaptation to preserve patients' outcome, but consistent data on the real efficacy of rehabilitative procedures are lacking, in particular concerning the rehabilitation effect on brain networks.

Therefore, this project focuses on the degree to which imaging measures of functional brain activity can give new hints on the effects of motor rehabilitative protocols in multiple sclerosis patients' performance. Particularly, the investigator's aim is to investigate the effects of upper limb rehabilitation, focused on hand motor function, and the correlation between motor performance and functional magnetic resonance data.

ELIGIBILITY:
Inclusion Criteria:

* Multiple sclerosis diagnosis according to McDonald criteria
* right handedness as assessed by the Edinburgh Handedness Inventory
* absence of relapses in the last three months
* mild or moderate sensorimotor impairment in one or both upper limbs as evaluated by means of the Medical Research Council scale (grade 3-4)

Exclusion Criteria:

* steroid-use or a worsening of the Expanded Disability Status Scale (EDSS) score in the last three months
* psychiatric disorders
* severe cognitive impairment
* magnetic resonance imaging contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2014-12-22 (Actual); Study Completion 2015-03-04 (Actual)

PRIMARY OUTCOMES:
Change in the time to perform the Nine Hole Peg Test (NHPT) | Baseline and 8 weeks
  The NHPT is a brief, standardized, quantitative test of upper extremity function, requiring participants to repeatedly place and then remove nine pegs into nine holes, one at a time, as quickly as possible.

SECONDARY OUTCOMES:
Score obtained at the Action Research Arm Test (ARAT) | Baseline and 8 weeks
  The Action Research Arm Test is an observational measure used to assess upper extremity performance (coordination, dexterity and functioning). The scale ranges from 0 to 57, with higher scores indicating better outcomes. Items are categorized into four subscales: grasp (score 0-18) , grip (0-12), pinch (0-18) and gross movement (0-9) which are arranged in order of decreasing difficulty, with the most difficult task examined first, followed by the least difficult task.
Grip and pinch strength | Baseline and 8 weeks
  Force applied by the hand and the fingers measured by means of specific dynamometers
Brain activity (blood-oxygenation-level dependent signal) | Baseline and 8 weeks
  Task-related brain activations assessed by means of functional magnetic resonance imaging during a finger-to-thumb opposition sequence

CONTACTS AND LOCATIONS:
Overall Officials: Marco Bove, Prof, Principal Investigator — Universita degli Studi di Genova

IPD SHARING:
Plan to Share IPD: No